CLINICAL TRIAL: NCT04326335
Title: Impact of Preoperative 3D Printed Stoma Placement on the Quality of Life of Ostomy Patients
Acronym: Stomie 3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD197-19
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-01

CONDITIONS: Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Felt-tip marking (Active Comparator)
  Interventions: Other: Felt-tip marking
- Felt-tip marking + 3D printed ostomy button (Experimental)
  Interventions: Other: Felt-tip marking + 3D printed ostomy button

INTERVENTIONS:
Other: Felt-tip marking — Marking the location of the future stoma with a felt pen
  Arms: Felt-tip marking
Other: Felt-tip marking + 3D printed ostomy button — Marking the location of the future stoma with a felt pen + 3D printed ostomy button placed on the future stoma location
  Arms: Felt-tip marking + 3D printed ostomy button

SUMMARY:
The making of an ostomy in patients is experienced as traumatic. The stoma changes body image, self-esteem and is responsible for increased anxiety. These changes affect the quality of life of patients. To reduce the negative impact of the stoma, patients are seen in preoperative consultation by the stoma nurses. This consultation allows to show the patients the appearance of a stoma (through a photograph), the equipment used and how it works.

In 2016, McKenna et al. showed the interest of marking (with felt pen) the ostomy site on the abdomen in preoperative. In this study, patients with preoperative marking had a higher post-operative quality of life score than patients without marking (p=0.03).

Quality of life was assessed using the STOMA-QOL score. This quality of life score is specific for ostomy patients. It assesses 4 dimensions: sleep, intimate relationships, relationships with family and close friends, relationships with people other than family and close friends. This questionnaire includes 20 questions and has been validated in 5 languages including French.

The aim of this pilot study is to evaluate the post-operative quality of life of ostomy patients who have benefited from a preoperative therapeutic education session with the placement of the 3D printed ostomy button versus felt-tip marking, during the 15 days prior to the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* First ileostomy with indication for temporary stoma placement,
* Patient with scheduled surgery,
* Patient who has the capacity to understand the protocol and has given consent to participate in the research,
* Patient with social security coverage.

Exclusion Criteria:

* Patient < 18 years old,
* Patient with an indication for placement of a permanent stoma,
* Emergency surgery patient,
* Patient who are pregnant, breastfeeding, or who have the potential to become pregnant without effective contraception,
* Patient under guardianship, curators or legal protection,
* Patient participating in another interventional clinical research protocol involving a drug or medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the post-operative quality of life of ostomy patients having benefited from preoperative therapeutic education sessions with 3D printed ostomy button placement versus felt marking. | 2 months post-discharge
  Total score on the Stoma-QOL (Quality-Of-Life) questionnaire The points obtained for each of the 20 questions are added together to obtain an overall score. This raw summary score per patient in the 20-80 range will be converted into a final score "0-100 score" where 0 indicates the worst Quality of Life and 100 the best Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Principal Investigator — Centre Hospitalier Departemental Vendee
Locations (1):
- Centre Hospitalier Departemental Vendee, La Roche-sur-Yon, France